CLINICAL TRIAL: NCT02718092
Title: Randomized Trial Comparing Fully Covered, Self Expanding Metal Stent (FCSEMS) and Plastic Stents for EUS- Guided Drainage of Walled -Off Necrosis (WON)
Brief Title: Comparing Fully Covered, Self Expanding Metal Stent (FCSEMS) and Plastic Stents for EUS- Guided Drainage of WON
Acronym: WON
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to pursue study
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jeffrey Easler, Assistant Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1512035809
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Walled-off Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Plastic Stent (Active Comparator): Three 7 Fr OR two 10 Fr Plastic Stents will be used
  Interventions: Device: Plastic Stent
- Axios FCSEMS (Active Comparator): 15 mm Axios Fully Covered Self Expanding Metal Stent
  Interventions: Device: Axios Fully Covered Self Expanding Metal Stent

INTERVENTIONS:
Device: Plastic Stent — Subjects who are randomized to this arm will receive a plastic stent
  Arms: Plastic Stent
Device: Axios Fully Covered Self Expanding Metal Stent — Subjects who are randomized to this arm will receive the Axios FCEMS
  Arms: Axios FCSEMS

SUMMARY:
This is a multi-center, single-blinded, randomized trial comparing AXIOS FCSEMS (Fully Covered Self Expanding Metal Stent) and plastic stents for EUS (Endoscopic Ultrasound)-guided management of infected and/or symptomatic WON (Walled Off Necrosis).

Patients will be randomized to either FCSEMS or plastic stents for EUS-guided drainage of WON in a 1:1 manner. Following EUS-guided drainage patients in both groups will be assessed pre- procedure, pre -discharge, weeks 1, 6 and months 3, 6, 12 and 24 months. Information will also be collected from any subsequent hospital admissions related to their walled-off necrosis.

DETAILED DESCRIPTION:
Consenting eligible patients will sign an IRB (Institutional Review Board)-approved, written informed consent to verify their willingness to participate in this study. Informed consent will be obtained on the day of their scheduled endoscopic drainage procedure and will occur at the time of consent to undergo the endoscopic drainage procedure (standard of care). Consent for the study will be obtained by one of the participating endoscopists and/or a research assistant. Subjects will receive a copy of the signed and dated informed consent document. Original informed consent documents will be maintained on-file at each participating center and will be made available for review upon request by coordinating center team or IRB, and/or any additional oversight organizations. A note may be made in the subject's hospital chart regarding participation in the research study. Once consented and enrolled into the trial, subjects will be issued a unique code to be used on data collection forms and other research records throughout the duration of the trial.

Preparation, Imaging and Endoscopic Procedures:

Patients on anti-platelet therapy or anticoagulation

1. Warfarin is to be stopped prior to the procedure per institutional guidelines..
2. Patients on heparin:

   1. Subcutaneous low molecular weight heparin (LMWH) is held for 12 hours and restarted the day after the procedure
   2. Intravenous heparin drip is stopped per institutional guideline prior to the procedure and restarted 12 hours after the drainage procedure
3. Aspirin can be continued until the day of the procedure
4. Clopidogrel and other anti-platelet agents are to be stopped per institutional guidelines prior to the procedure and restarted the day after the procedure. In patients with placement of drug-eluting stents within one year, the risk of cessation of clopidogrel will have to be weighed against the risk of bleeding during the drainage procedure. In that case, cardiology may be consulted so that the best course of action can be taken.

Imaging prior to EUS-guided drainage

1. MRI (Magnetic Resonance Imaging) / MRCP (Magnetic Resonance Cholangiopancreatography) with gadolinium will be performed in all patients to assess the WON. In patients with contraindications to MRI, a CECT ( Contrast Enhanced, Computed Tomography) abdomen/pelvis will be obtained instead. In patients with contraindication to both MRI/MRCP and intravenous iodinated contrast (such as history of anaphylactic reaction to iodinated contrast agents or renal impairment with eGFR < 30 mL/min/1.73m2), a non-contrast enhanced CT will be performed. All imaging will be interpreted by the designated GI/abdominal radiologist at each participating center and also by an appointed multidisciplinary panel to determine suitability for inclusion in the study.
2. In addition to MRI/CT, EUS will be utilized at the time of the drainage procedure in the final determination of the percentage of pancreatic necrosis.
3. ERCP (Endoscopic Retrograde Cholangiopancreatography) will not be mandatory prior to EUS-guided drainage as the incidence of disconnected pancreatic duct syndrome (DPDS) is high and the placement of a pancreatic duct stent is unlikely to be helpful in this case.

Endoscopic Drainage

1. Intravenous antibiotic (e.g. ciprofloxacin, levofloxaen or augmentin) is administered on the day of the procedure. Oral antibiotics will be continued for ten days following drainage.
2. All procedures are performed under general anesthesia.
3. One drainage site is created in all WON, regardless of size or stent type.
4. Percutaneous drainage is not undertaken prior to EUS-guided drainage.
5. Insertion of plastic stents:

   1. WON is first identified using EUS, and punctured using a 19G needle. 20cc of the pancreatic fluid is aspirated and sent for CEA, amylase, cell count, gram stain and culture with sensitivities. A 0.025 or 0.035 inch guidewire is inserted into the WON through the FNA (Fine Needle Aspirate) needle. A transmural tract is created using an ERCP catheter (with the use of a needle knife catheter ± cautery if needed), and then dilated using a 12-13.5-15mm CRE balloon to a maximum size of 15mm if technically possible. Three 7Fr OR two 10Fr plastic stents are inserted through the transmural tract into the WON cavity.
   2. A nasocystic catheter is placed into the WON through the plastic stent and irrigated every six hours using 250 cc of normal saline for 48 hours. The patient will remain in-patient for irrigation of the nasocystic catheter. If an attempt at nasocystic catheter fails the endoscopist will attempt to lavage the cystic cavity with 2L of saline at that time with 2L of sterile water.
   3. If placement of the nasocystic catheter and lavage fails and/or is not deemed to be safe, this will be documented and no further action is taken.
6. Insertion of AXIOS FCSEMS:

   1. WON is first identified using EUS and punctured using a 19G needle. Enough fluid is aspirated to send for CEA, amylase, cell count, gram stain and culture with sensitivities.
   2. A 0.025 or 0.035 inch guidewire is inserted into the WON through the FNA needle. A transmural tract is created using ERCP dilation catheters or electrocautery devices ( needle knife catheter or Hot Axios cautery if needed) as described below. The catheter-based stent delivery system with a 15mm AXIOS stent mounted onto it is inserted into the endoscope, and introduced into the WON cavity either: 1) after dilation with endoscopic dilators (4-5-7 French/5-7-10 French push dilators, 4mm, or 6mm balloons) or 2) using electrocautery mounted on the stent system ("Hot Axios"). The stent should be positioned so that it lies within both the WON and enteric lumen. The stent is then deployed so that one flange of the stent is located within the WON cavity and the other flange is located within the enteric lumen. The Axios stent is then dilated to at least 13.5-15mm following deployment using a 12-15mm balloon.
   3. An attempt at irrigation/lavage of the WON cavity in the endoscopy unit immediately following stent deployment using 2L of normal saline should be performed. This can be done using a forward viewing gastroscope or endoscopic accessories (push dilation catheters, balloon catheters etc.).
7. Direct endoscopic necrosectomy will not be performed in the same session as the initial stent placement.
8. The following information is collected at the time of initial endoscopic procedure:

   1. Location and size of collection by EUS measurements (two perpendicular measurements)
   2. Intraprocedure complications (such as bleeding, pneumoperitoneum, perforation, hemodynamic instability)
   3. Procedure duration

   i. Initial procedure (start time: advancement of the endoscope into the patient; end time: withdrawal of the echoendoscope, gastroscope or duodenoscope from the patient at the end of the procedure)

Follow-up Procedures:

Post-procedure management:

1. Oral antibiotics will be administered for a total of ten days pending the results of fluid gram stain and culture. Antimicrobial therapy will thereafter be altered based on fluid culture results as indicated.
2. All patients will be admitted for no less than 48 hours for observation after the index endoscopic procedure.
3. Enteral nutrition will be commenced within 48 hours of the procedure via nasogastric tube, PEG-J (Percutaneous endoscopic gastrostomy tube with a jejunal extension), nasojejunal tube or surgical/endoscopic jejunostomy or through the prompt transition to oral diet unless contraindicated. Route of enteral nutrition support will be determined by the treating physician.
4. In the plastic stent group, the WON is irrigated using 250cc of normal saline every six hours for total duration of 48 hours. The nasocystic catheter is removed after 48 hours.

At 48-96 hours post-procedure:

1. MRI/CECT (if contraindication to MRI) is obtained if any of the following criteria are met:

   a. Persistent symptoms of abdominal pain, gastric outlet obstruction and/or failure to advance diet b. Ongoing SIRS (Systemic Inflammatory Response Syndrome) /Sepsis c. Persistent organ failure
2. If the above repeat MRI/CECT fail to show resolution of WON (defined as ≥50% decrease in volume), a repeat intervention is performed
3. The type of repeat intervention performed is to be determined by the treating physician and can include:

   1. Direct endoscopic necrosectomy (DEN) in unilocular collection with significant solid component
   2. Creation of a second drainage site and/or DEN in multi-loculated/large collection without a significant solid component
   3. Placement of interventional radiology-guided percutaneous drain in collections not accessible via the stomach/duodenum
4. Repeat interventions are performed at a frequency determined by the treating physician until the volume of WON has decreased ≥ 50% with clinical improvement, up to maximum of three sessions.
5. If there is still inadequate response to treatment (as defined above) after three endoscopic transmural drainage procedures using the designated stent type (i.e. procedure #1=stent insertion, procedure #2-3= insertion of more stents into a second drainage site ± direct endoscopic necrosectomy ± percutaneous drain insertion), the patient is defined as "endoscopic treatment failure". These patients will be referred for minimally invasive surgical debridement of WON.
6. Procedures #2 and 3 will also be undertaken as described above for patients returning to the hospital in the period following discharge after index procedure.

Pre-discharge:

Following information is obtained prior to discharge:

1. Symptoms:

   a. Pain b. Nausea/vomiting c. Malaise d. Oral intake (liquid diet, solid diet, duration of tolerance to po intake)
2. Adverse events
3. Need for repeat endoscopic procedures: percutaneous drain placement, surgery
4. VAS pain score

At Week 1: (+ or- 2 days)

Telephone calls are made to all patients to collect the following information:

1. Symptoms
2. Adverse events
3. VAS pain score
4. SF-36

At Week 6: (+ or -7 days)

1. Repeat MRI/MRCP with gadolinium (or CECT if MRI contraindicated) is performed to reassess the size of WON and to look for disconnected pancreatic duct syndrome (DPDS):

   1. If DPDS is present on MRI/CT, no ERCP is done
   2. If DPDS if not present on MRI/CT, ERCP is performed the following day to confirm patency of the pancreatic duct. If a partial pancreatic duct leak is present on ERCP, a transpapillary stent is placed during the same endoscopic session. Repeat ERCP with stent exchange is to be performed at the discretion of the endoscopist.
2. If the WON is < 10% of its original size (defined as treatment success),:

   a. All transmural stents are removed if the main pancreatic duct (MPD) is intact.

   b. If the MPD is disconnected, all but one plastic stent is removed. A single double pigtail plastic stent will be left in place indefinitely. In patients with FCSEMS and DPDS, the metal stent is removed and a single 7Fr double pigtail plastic stent is placed instead and left in place indefinitely. FCSEMS is replaced with double pigtail plastic stents in this group as thus far the long-term sequelae of inserted AXIOS stents are not known, including the risk of stent migration.
3. If at or during the first 6 weeks after the initial drainage procedure, there no resolution of WON and/or persistent symptoms repeat interventions are performed.
4. The type of repeat intervention performed is to be determined by the treating physician with suggestions listed below. These can include:

   1. Direct endoscopic necrosectomy (DEN) in unilocular collection with significant solid component
   2. Creation of a second drainage site and/or DEN in multi-loculated/large collection without a significant solid component
   3. Placement of interventional radiology-guided percutaneous drain in collections not accessible via the stomach/duodenum
   4. Referral for minimally invasive surgical debridement of WON. Surgical intervention should be considered in patients with significant, ongoing debilitating symptoms.
5. MRI/MRCP is then again repeated 6 weeks following the second round of drainage procedures to check for WON resolution
6. If there is no resolution of WON following the second endoscopic drainage, repeat intervention(s) as outlined in 4) is performed.
7. MRI/MRCP is then again repeated 6 weeks following the third drainage to check until WON resolution
8. If there is no resolution of WON following the third endoscopic drainage, the patient must be referred for minimally invasive surgical necrosectomy
9. Documentation of symptoms or adverse events
10. Admissions
11. VAS score
12. SF-36 questionnaire Any subsequent admissions (related to the Walled Off- Necrosis)

The following information will be collected in patients hospitalized with recurrent symptoms:

1. Symptoms
2. Adverse events
3. VAS pain score or admission recorded pain score if at any outside hospital
4. Need for subsequent endoscopic, percutaneous or surgical procedures for WON
5. Duration of Hospital stay

At Month 3, 6, 12, 24: (+ or - 14 days)

Telephone calls are made to all patients to gather information on the outcome measures:

1. Documentation of symptoms or adverse events
2. Admissions
3. VAS score

1) SF-36 questionnaire ( Months 6, 12 and 24 only)

5) MRI/MRCP or CT scan at 6 months in patients with initial treatment success to determine rate of WON recurrence

ELIGIBILITY:
Inclusion Criteria:

1. WON diagnosed on contrast-enhanced dual phase CT abdomen/pelvis (CECT) or MRI with gadolinium (seen as a fluid collection in the setting of documented pancreatic necrosis that contains necrotic material and encased within a well-defined tissue layer)
2. All WON centered within the pancreatic/peri-pancreatic space not requiring percutaneous drainage, ≥ 6cm, located within 2cm of the enteric wall, not extending into the flanks or pelvis
3. WON with single loculation, with no extension into the flanks, pelvis or into the root of the small bowel mesentery. Collections should have an estimated solid component of = or >25% based on cross sectional imaging and/or endosonographic evaluation of the collection at the time of study procedure.
4. Suspected/confirmed infected WON (defined as temp ≥ 100.5°F, serum WBC ≥ 15x199/L, positive blood cultures or positive Gram stain/culture of aspirated necrotic material) and/or
5. Symptomatic WON (defined as abdominal pain, gastric/intestinal/biliary outlet obstruction resulting in nausea, vomiting, early satiety, jaundice, or persistent malaise) at a time interval of ≥ 4 weeks from attack of acute pancreatitis complicated by pancreatic necrosis
6. Documented history of acute or chronic pancreatitis

   a) Acute pancreatitis is diagnosed if 2 of the following 3 criteria are met: i) Abdominal pain characteristic of acute pancreatitis ii) Serum lipase/amylase ≥ x3 upper limit of normal iii) Characteristic radiological findings of acute pancreatitis on CECT/MRI/US abdomen, such as homogeneous enhancement of pancreatic parenchyma, standing of peripancreatic fat (1) b) Chronic pancreatitis is diagnosed if characteristic radiological changes are seen on CT/MRI with MRCP (such as pancreatic atrophy, dilated pancreatic duct, pancreatic calcification) (11) or EUS (≥5/9 of Rosement criteria) (12)
7. Able to undergo general anesthesia

Exclusion Criteria:

1. Age < 18 years
2. Unable to obtain consent for the procedure
3. Pregnancy
4. Irreversible coagulopathy: INR > 1.5, platelets < 50 x 109/L
5. Use of anticoagulants that cannot be discontinued for the procedure
6. Unable to tolerate general anesthesia
7. WON with ≥ 3 loculations
8. WON that is not accessible for EUS-guided drainage
9. Percutaneous drainage of WON is required or performed prior to EUS-guided drainage
10. Prior endoscopic, percutaneous or surgical drainage procedure(s) for pancreatic/peri-pancreatic fluid collections.
11. Contraindication to endoscopic drainage: Gastrectomy with Billroth II, gastric bariatric surgery, prior pancreatic surgery, prior esophagectomy, cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Short term efficacy as measured by interval decrease in size in WON (Walled Off Necrosis) collection to 10% of the pre-treatment volume as measured in centimeters^3. | 6 weeks
  Hypothesis: Short term efficacy for radiographic resolution of symptomatic walled off necrosis. Diameter of the collection on MRI/CT axial and coronal imaging sections will be used to calculate volume in centimeters ^3.
Short term efficacy as measured with improvement in symptoms using Visual Analog Scale (VAS) | 6 Weeks
  Visual Analog Pain Scale Ranges. 0= No pain Ever to 10= Worst Pain. Visual faces demonstrate increased unhappiness as the numbers rise
Short term efficacy as measured with improvement in symptoms using the SF-36 questionnaire scale | 6 weeks
  SF-36 is a 36 question, patient reported survey of patient health. It is a measure of health status.
Long term efficacy as measured by interval decrease in size in WON collection to 10% of the pre-treatment volume as measured in centimeters^3. | 24 Months
  Hypothesis: Long term efficacy for radiographic resolution of symptomatic walled off necrosis. Diameter of the collection on MRI/CT axial and coronal imaging sections will be used to calculate volume in centimeters ^3.
Long term efficacy as measured with improvement in symptoms using Visual Analog Scale (VAS) | 24 Months
  Visual Analog Pain Scale Ranges. 0= No pain Ever to 10= Worst Pain. Visual faces demonstrate increased unhappiness as the numbers rise
Long term efficacy as measured with improvement in symptoms using the SF-36 questionnaire scale | 24 Months
  SF-36 is a 36 question, patient reported survey of patient health. It is a measure of health status.

SECONDARY OUTCOMES:
Using the perspective of the payer, obtain and extrapolate cost data to compare direct healthcare costs | 24 months from stent insertion.
  Investigators plan to collect data on "actual" healthcare expenses for hospital, facility and physician charges in the form of CPT and ICD-10 data generated during the management of walled of necrosis accrued during the study period at the time of and following stent insertion for patients enrolled in the study.
  "Hypothetical costs" will also be extrapolated by average price unit for procedures, equipment, anesthesia costs, length of inpatient stay and level of inpatient care.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Easler, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No